CLINICAL TRIAL: NCT05622188
Title: HEAT Stress Detection From Personally STandARdized Heat Strain Measurements - The HEATSTAR Pilot Trial
Brief Title: The Detection of Heat Stress by Assessing Individual Body Responses to Heat (Heat Strain) in Young and Healthy Non-athlete Participants
Acronym: HEATSTAR
Status: Completed | Type: Observational
Sponsor: ETH Zurich (Other)
Collaborators: Swiss Federal Office of Sports (BASPO) (Unknown); University of Zurich (Other); Center for Chronobiology, Psychiatric University Clinics, Basel (Unknown); epyMetrics (Unknown); Innosuisse - Swiss Innovation Agency (Other); Swiss Federal Railways (Unknown)
Responsible Party: Principal Investigator, Noe Brasier, Principal Investigator, ETH Zurich
Other Study IDs: EKNZ ID: 2022 - 01325
Record Dates: First submitted 2022-11-11; First posted 2022-11-18 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Heat Stress
Keywords: Heat Strain; Wearable; Sweat Analysis
MeSH Terms: conditions — Heat Stress Disorders | interventions — Physical Exertion

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy participants: Age of the participants is between 18-40 years, females and males equally distributed
  Interventions: Other: Elevated ambient heat; Other: Elevated relative humidity; Other: Exertion

INTERVENTIONS:
Other: Elevated ambient heat — Temporary exposure to increased ambient temperature +10°C (the effect of the intervention is fully and spontaneously reversible)
Other: Elevated relative humidity — Temporary exposure to increased ambient relative humidity +40% (max. 90%) (the effect of the intervention is fully and spontaneously reversible)
Other: Exertion — Temporary exertion on an ergometer (1W/kg body weight) (the effect of the intervention is fully and spontaneously reversible)

SUMMARY:
• This study investigates and compares the within and in-between variances of the body responses to different heat stressors in a controlled lab-setting. The participants will be exposed to different heat sources while a variety of physiological heat strain reactions such as heartrate, sweat rate, and core body temperature are recorded using on- and in-body devices. For the participant monitoring during the study, medical grade devices such as a certified ECG and a swallowable sensor-pill to continuously monitor the core body temperature will be applied. A one-for-all wearable device is additionally applied for physiological validation. Further, sweat will be collected to assess (i) the local sweat rate and (ii) the appearance of different heat stress associated molecular markers in this non-invasively collectable biofluid. As a secondary aim, a model will be developed that will enable to predict the different heat stress sources out of the heat strain measurements.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participant, able to give consent
* Age 18-40 years
* Non-athlete (<4h sport/week)
* BMI<30 (non-obese)
* German speaking, or fluent in German

Exclusion Criteria:

* Pregnancy (urine pregnancy test), and breastfeeding
* Regular medication intake (excluding birth control pill)
* Intake of drugs and/or daily alcohol consumption
* Fever or symptoms of an acute infection (cough, shortness of breath, sore throat, taste loss)
* Active smoking or history of smoking <9 months ago
* Mobility impairment
* Traveled (<1 month ago) to a warm/hot temperature zone and stayed for >6 days
* Any chronic conditions such as: high blood pressure, diabetes mellitus, immuno-deficiencies, sweat disorders such as anhidrosis
* Color blindness (STROOP test)
* Weight <40 kg (e-Celsius pill)
* Diverticulum or obstructions of the gastrointestinal tract (including motility disorders, swallowing disorders) as well as major abdominal surgery (e-Celsius pill)
* Need of exposure to strong electromagnetic fields during study participation, above all MRI examinations (e-Celsius pill)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants will be recruited through Swiss Universities and Swiss Universities of Applied Science. The institutions host a broad range of students that are likely to match the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2022-11-02 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-02-10 (Actual)

PRIMARY OUTCOMES:
The within and between subject heat strain marker variability in relation to specific heat stress sources (ambient heat, ambient humidity, exertion, and clothing) | Max. 7 days
  The primary endpoint is the within- and between- subject heat strain marker variability of HR, CBT, WSR, and LSR in relation to various heat stress sources (increased ambient temperature, increased relative humidity, and exertion, all without and with additional clothing.

SECONDARY OUTCOMES:
Accuracy to detect the specific heat stress source (such as ambient heat, relative humidity) from different on- and in-body measurements | Max. 7 days
  The models for the primary endpoints will be extended to explore the relationships between heat strain parameters, heat stress sources, as well as personal characteristics. Additionally, prediction of heat stress source will be explored.
Assessment of short-term heart rate variability in context to each heat stressor. | Max. 7 days
  Short-term HRV with a repeating time frame of 5min. Root mean square of successive RR interval (RMSSD; in [ms]) and the Standard-deviation of RR intervals (SDRR; in [ms]) will be computed with respect to each heat stress source.
Temperature [°C] and relative humidity [%] of the microenvironment as an additional source of information for patterns to detect heat stressors | Max. 7 days
  Features of temperature [°C] and relative humidity [%] of the microenvironment as additional model predictors.

OTHER OUTCOMES:
The relation between cognitive assessment and skin temperature | Max. 7 days
  Correlation between subjective heat comfort (Visual Analog Scale, where +1 is comfortable and +4 is very uncomfortable) and baseline differential stress inventory (causes of stress, symptoms of stress, coping, stress stabilization) in relation to skin temperature [°C]
The relation between STROOP assessment and different heat stressors | Max. 7 days
  Correlation between changes in the STROOP assessment outcome (number of errors and time of decision [ms], between beginning and end of heat stress exposure) in context to the various heat stress sources, skin temperature, and thermal comfort.
Novel Sweat Biomarkers for heat stress detection | Max. 7 days
  Descriptive statistics for novel non-invasive biomarkers from sweat analysis with respect to heat stress source, including between- and within-subject variability
Recording heat strain parameters with an all-for-one device | Max. 7 days
  The 'reliability' (missing data per minute ([%]) and the 'accuracy' (HR [bpm] with 95% confidence intervals), CBT (in [°C] with 95% confidence intervals), and local sweat rate measurements (in [g/h] with 95% confidence intervals) of the wearable device in recording vital parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Noé Brasier, MD, Principal Investigator — ETH Zurich
Locations (1):
- ETH Zurich, Zurich, Andere (Nicht USA-Länder), Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Watts N, Amann M, Ayeb-Karlsson S, Belesova K, Bouley T, Boykoff M, Byass P, Cai W, Campbell-Lendrum D, Chambers J, Cox PM, Daly M, Dasandi N, Davies M, Depledge M, Depoux A, Dominguez-Salas P, Drummond P, Ekins P, Flahault A, Frumkin H, Georgeson L, Ghanei M, Grace D, Graham H, Grojsman R, Haines A, Hamilton I, Hartinger S, Johnson A, Kelman I, Kiesewetter G, Kniveton D, Liang L, Lott M, Lowe R, Mace G, Odhiambo Sewe M, Maslin M, Mikhaylov S, Milner J, Latifi AM, Moradi-Lakeh M, Morrissey K, Murray K, Neville T, Nilsson M, Oreszczyn T, Owfi F, Pencheon D, Pye S, Rabbaniha M, Robinson E, Rocklov J, Schutte S, Shumake-Guillemot J, Steinbach R, Tabatabaei M, Wheeler N, Wilkinson P, Gong P, Montgomery H, Costello A. The Lancet Countdown on health and climate change: from 25 years of inaction to a global transformation for public health. Lancet. 2018 Feb 10;391(10120):581-630. doi: 10.1016/S0140-6736(17)32464-9. Epub 2017 Oct 30. No abstract available. PMID 29096948
- [Background] Varghese BM, Hansen A, Bi P, Pisaniello D. Are workers at risk of occupational injuries due to heat exposure? A comprehensive literature review. Safety Science. 2018;110:380-92.
- [Background] Davey SL, Downie V, Griggs K, Havenith G. The physiological strain index does not reliably identify individuals at risk of reaching a thermal tolerance limit. Eur J Appl Physiol. 2021 Jun;121(6):1701-1713. doi: 10.1007/s00421-021-04642-3. Epub 2021 Mar 7. PMID 33677693
- [Background] Nunes MJ, Cordas CM, Moura JJG, Noronha JP, Branco LC. Screening of Potential Stress Biomarkers in Sweat Associated with Sports Training. Sports Med Open. 2021 Jan 22;7(1):8. doi: 10.1186/s40798-020-00294-3. PMID 33481103
- [Background] Flores M, Glusman G, Brogaard K, Price ND, Hood L. P4 medicine: how systems medicine will transform the healthcare sector and society. Per Med. 2013;10(6):565-576. doi: 10.2217/pme.13.57. PMID 25342952